CLINICAL TRIAL: NCT02371915
Title: Addressing Rural and Remote Access Disparities for Patients With Inflammatory Arthritis Through Telehealth/Videoconferencing and Innovative Inter-professional Care Models
Brief Title: Interprofessional Care Models Using Videoconferencing for Patients With Inflammatory Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Initiative for Outcomes in Rheumatology Care (Other)
Responsible Party: Principal Investigator, Regina M. Taylor-Gjevre, Professor of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-176
Record Dates: First submitted 2014-12-08; First posted 2015-02-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Inflammatory Arthritis
Keywords: Rural access; Telehealth
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videoconference follow-up (Experimental): These subjects will remain in or near their home communities for rheumatology follow-up visits. Follow-up visits will occur via telehealth/videoconferencing, with a physiotherapist present, performing the in-person assessment, supported by the rheumatologist via videoconference.
  Interventions: Other: Videoconference follow-up
- Control (No Intervention): These subjects will continue to travel into Saskatoon for the rheumatology visits, as they normally would for routine follow-up visits with their rheumatologist.

INTERVENTIONS:
Other: Videoconference follow-up — Rheumatology visits to take place video videoconference with a physiotherapist present
  Arms: Videoconference follow-up

SUMMARY:
This project will be conducted in two phases. Phase 1: RA patients will be recruited to participate in five repeated examinations occurring in one day to compare between and within specialties, ensuring reasonable equivalency of examination findings. Phase 2: RA patients living > 100 km from Saskatoon will be randomized to the intervention or control group, with both groups having three follow-up appointments in 3-month intervals. The intervention group will be evaluated by a physiotherapist supported by a rheumatologist through videoconferencing, while the control group will continue to travel to Saskatoon for follow-up care.

DETAILED DESCRIPTION:
Part A: Validation Study This study involves inter-professional care with rural-based physical therapists and urban-based rheumatologists, it will be a valuable first step to validate comparability of the physical examination. We shall compare physical examination accuracy between and within examiner disciplines. Examiners will include the three rheumatologist study investigators and three participating physical therapists with additional training in inflammatory rheumatic diseases and experienced in musculoskeletal assessment.

Procedures: All examiners will undergo a standardized review of examination techniques and documentation prior to participating.

Comparison groups will be:

1. Rheumatologist A. to Rheumatologist B.
2. Physiotherapist A. to Physiotherapist B.
3. Rheumatologist A/B to Physiotherapist C/teleconferenced Rheumatologist C. We will use web-based videoconferencing software. This desktop-based solution is currently being piloted by Telehealth Saskatchewan and is used extensively in Ontario. This technology satisfies Health Information Protection Act (HIPA) as well as the Saskatchewan privacy and security concerns. An examining room with telehealth/videoconference equipment will be available for patient distance examination for comparison group C as listed above. The rheumatologist will be in a physically separate room with viewing equipment in a mock distance evaluation. The proposed study will be conducted in cooperation with the Canadian Centre for Health and Safety in Agriculture (CCHSA) within the ≈1350 m2 National Agricultural-Industrial Hygiene Laboratory. Clinical visits will be conducted at the CCHSA.

Part B: Randomized Controlled Rheumatoid Arthritis Care Delivery Model Trial Randomization: Participating patients will be randomly allocated to two arms, either to be followed by telehealth/videoconferencing in or near their home community or to continue traveling to their Saskatoon rheumatology clinic.

Intervention: One study arm will be followed in traditional rheumatology clinic (in-person examining rheumatologist). The second study arm will be followed by telehealth/videoconferencing. Patients in the telehealth/videoconferencing arm will be examined by a rural-based physical therapist who will report exam findings during telehealth review with the urban-based rheumatologist. Follow-up visits will be every three months in both arms. All patients will complete standardized history/data-collection forms. Patients will be followed in their respective study arms for nine months, and then will be evaluated in-person in rheumatology clinic for final face-to-face disease activity evaluation.

ELIGIBILITY:
Inclusion Criteria:

Part A: Patients with established rheumatologist diagnosed RA attending rheumatology clinic at Royal University Hospital, (Saskatoon) and providing informed consent, will be recruited.

Part B: As the target population for future telehealth/VC utilization will be patients living outside the urban centers, participants will be similarly selected. Inclusion criteria will be: age over 18 years, ability to provide informed consent, place of residence 100 kilometers or more outside of Saskatoon, and rheumatologist established diagnosis of rheumatoid arthritis.

Exclusion Criteria:

Exclusion criteria will include participation in the earlier validation study (Part A).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity Score-28 (DAS-28) | at 3 month intervals over nine months

SECONDARY OUTCOMES:
Change in European Quality of Life - 5 Dimensions(EQ-5D) | at 3 month intervals over nine months
Change in Epworth Sleepiness Scale | at 3 month intervals over nine months
Change in Healthcare Use | at 3 month intervals over nine months
Change in Modified Health Assessment Questionnaire (MHAQ) | at 3 month intervals over nine months
Change in Work Productivity and Activity Impairment Questionnaire (WPAI) | at 3 month intervals over nine months
Change in International Physical Activity Questionnaire (IPAQ) | at 3 month intervals over nine months
Change in Rheumatoid Arthritis Disease Activity Index (RADAI) | at 3 month intervals over nine months

CONTACTS AND LOCATIONS:
Overall Officials: Regina Taylor-Gjevre, MD, Principal Investigator — Univsersity of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No